CLINICAL TRIAL: NCT02286531
Title: Evaluation de O-(2-[18F]-Fluoroethyl)-L-Tyrosine (or FET), a New Tracer PET (Positron Emission Tomography) , in the Diagnosis of Low Grade Glioma
Brief Title: Evaluation de O-(2-[18F]-Fluoroethyl)-L-Tyrosine, a New Tracer PET, in the Diagnosis of Low Grade Glioma
Acronym: PET-FETII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08 111 01
Record Dates: First submitted 2014-11-04; First posted 2014-11-10 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Low Grade Glioma
Keywords: : Low grade glioma; PET; FET; MRI; Standardized uptake value
MeSH Terms: interventions — O-(2-fluoroethyl)tyrosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FET imaging (Experimental): FET Imaging. Patient 0.1 mCi / kg (maximum 185 MBq) of FET with 'O-(2[18F]FLUOROETHYL)-L-TYROSINE' will be injected through the venous catheter. At the same time, will trigger a PET 3D dynamic acquisition of 60 minutes (5 pictures 1 minute and 11 images of 5 minutes)
  Interventions: Drug: O-(2[18F]FLUOROETHYL)-L-TYROSINE

INTERVENTIONS:
Drug: O-(2[18F]FLUOROETHYL)-L-TYROSINE — Patient 0.1 mCi / kg (maximum 185 MBq) of FET will be injected through the venous catheter. At the same time, will trigger a PET 3D dynamic acquisition of 60 minutes (5 pictures 1 minute and 11 images of 5 minutes)
  Other Names: FET imaging

SUMMARY:
Determine the overall discriminatory ability of FET PET in the diagnosis of glioma grade II (referring to the current diagnostic gold standard represented by the histopathology exam of a tumor sample).

DETAILED DESCRIPTION:
Low-grade glioma is a malignant tumor of young adults (12.5% of gliomas, incidence of 0.99 / 100,000). Median survival, linked to anaplastic transformation is estimated between 7 and 10 years, with great individual variability in the rate of evolution. The morphological MRI, standard assessment tool at present, suffers from many limitations, especially concerning the positive diagnosis, the targeting of surgical biopsies and tumor delineation which is essential to treatment The study design is a validation study of a new diagnostic procedure. This study is prospective, no randomized, multicenter involving 10 centers (Toulouse University Hospital, Caen, Tours, AP-HP Pitie Salpetriere, Lille, Angers, Rennes, Nîmes, Nantes and Nancy). Will be eligible patients in whom the diagnosis of grade II glioma is suspected according to clinical data and MRI, after evaluation and multidisciplinary meeting at which histological confirmation is scheduled within a maximum period of one month.

FET PET scans will be performed before any procedure or surgical treatment and the data will be merged with MRI. The gold standard is histological examination or biopsy material, or complete resection of the tumor. A minimum of three biopsies per patient will be realized. The pathologist will not see the results of PET-FET 100 patients will be enrolled over a period of 5 years. The area under the curve will be determined on a non-parametric for each increase in the value of PET-FET at near 10th. The sensitivities, specificities, positive predictive values will be estimated with confidence intervals at 95%. Factors to be considered in the analysis, the intrasubject variability related to the fact that several positive and negative results are found for each subject included. The concordance between the data-FET PET and MRI will be sought.

The expected benefits are a better diagnostic ability of PET-FET which results in a specific targeting of biopsies with fewer tests to false negatives and false positives, thus a better diagnostic yield of this invasive procedure. Furthermore, the characteristics of this test applied to all of the tumor may help to better define the limit between healthy and tumor areas and thus reduce the radiation fields to the volumes strictly necessary. These volumes are currently defined on the results of the only morphological MRI and can be further clarified

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years

* Diagnosis of glioma grade II referred on clinical and MRI morphologic
* Realization of a brain MRI in preoperative condition of neuronavigation (MRI sequences including axial T2, Flair, T1, T1 with gadolinium) in a within 1 month with FET PET.
* Histological examination scheduled within one month with FET PET by resection (complete or partial) or by biopsy
* Patients who signed informed consent
* No against-indication for PET
* No against-indications to MRI

Exclusion Criteria:

* Grade II glioma who have received specific treatment with radiotherapy and or chemotherapy.
* Pregnant or breastfeeding women.
* Weight greater than 120 Kg
* against-indication to PET
* against- indication gadolinium
* Possible side effects to MRI (magnetic foreign bodies, pacemaker, congestive severe renal).)
* Patient under guardianship
* No coverage by social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Determine the overall discriminating capacity of FET-PET in the diagnosis of glioma grade II (referring to current diagnostic gold standard represented by the histopathological examination of a tumor sample). | TEP and MRI Imagy 1 month before surgery

SECONDARY OUTCOMES:
- Determine the threshold with the highest positive likelihood ratio. - Determine the threshold with the highest positive likelihood ratio. | 1 month before surgery
Assess the concordance of the data-FET PET and MRI morphological data reported to histological diagnostic | 1 month before surgery
Evaluate the positive and negative predictive value of this threshold in order to improve the delineation of the tumor area | 1 month before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Payoux, MD PHD, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - CHU de CAEN, Caen
  - Hôpital de la Pitié Salpétrière, Paris
  - UHToulouse, Toulouse